CLINICAL TRIAL: NCT03235193
Title: Prediction of Severe Sepsis Using a Machine Learning Algorithm
Brief Title: Predictive algoRithm for EValuation and Intervention in SEpsis
Acronym: PREVISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dascena (Industry)
Collaborators: Cabell Huntington Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: 1097090-1
Record Dates: First submitted 2017-07-27; First posted 2017-08-01 (Actual); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Sepsis; Septic Shock; Severe Sepsis
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- With InSight (Experimental): Healthcare provider receives an alert from InSight for patients trending towards severe sepsis. Healthcare provider also receives information from the severe sepsis detector in the CHH electronic health record.
  Interventions: Other: Severe Sepsis Prediction; Other: Severe Sepsis Detection
- Without Insight (Active Comparator): Healthcare provider does not receive any alerts from InSight. Healthcare provider receives information from the severe sepsis detector in the CHH electronic health record.
  Interventions: Other: Severe Sepsis Detection

INTERVENTIONS:
Other: Severe Sepsis Prediction — Upon receiving an InSight alert, healthcare provider follows standard practices in assessing possible (severe) sepsis and intervening accordingly.
  Arms: With InSight
Other: Severe Sepsis Detection — Upon receiving information from the severe sepsis detector in the CHH electronic health record, healthcare provider follows standard practices in assessing possible (severe) sepsis and intervening accordingly.

SUMMARY:
In this prospective study, the ability of a machine learning algorithm to predict sepsis and influence clinical outcomes, will be investigated at Cabell Huntington Hospital (CHH).

ELIGIBILITY:
Inclusion Criteria:

* All adult patients visiting the emergency department, or admitted to the participating intensive care unit (ICU) wards of Cabell Huntington Hospital will be eligible.

Exclusion Criteria:

* All patients younger than 18 years of age will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2296 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality | Through study completion, an average of 30 days

SECONDARY OUTCOMES:
Hospital length of stay | Through study completion, an average of 30 days

OTHER OUTCOMES:
Hospital readmission | Through study completion, an average of 30 days
ICU length of stay | Through study completion, an average of 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Hoyt Burdick, Principal Investigator — Cabell Huntington Hospital
Locations (1):
- Cabell Huntington Hospital, Huntington, West Virginia, United States

REFERENCES:
- [Background] Calvert J, Desautels T, Chettipally U, Barton C, Hoffman J, Jay M, Mao Q, Mohamadlou H, Das R. High-performance detection and early prediction of septic shock for alcohol-use disorder patients. Ann Med Surg (Lond). 2016 May 10;8:50-5. doi: 10.1016/j.amsu.2016.04.023. eCollection 2016 Jun. PMID 27489621
- [Background] Calvert JS, Price DA, Chettipally UK, Barton CW, Feldman MD, Hoffman JL, Jay M, Das R. A computational approach to early sepsis detection. Comput Biol Med. 2016 Jul 1;74:69-73. doi: 10.1016/j.compbiomed.2016.05.003. Epub 2016 May 12. PMID 27208704
- [Background] Desautels T, Calvert J, Hoffman J, Jay M, Kerem Y, Shieh L, Shimabukuro D, Chettipally U, Feldman MD, Barton C, Wales DJ, Das R. Prediction of Sepsis in the Intensive Care Unit With Minimal Electronic Health Record Data: A Machine Learning Approach. JMIR Med Inform. 2016 Sep 30;4(3):e28. doi: 10.2196/medinform.5909. PMID 27694098